CLINICAL TRIAL: NCT03476733
Title: Incidence and Risk Factor of Drug Related Problem Detected in Inpatient
Acronym: DRPINPAT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0135
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Drug Related Problem
Keywords: Drug related problem; inpatient; Medication Error; Clinical Pharmacist
MeSH Terms: interventions — Inosine Monophosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient with drug related problem: patient with drug related problem
  Interventions: Other: Detection of drug related problem in inpatient
- patient without drug related problem: patient without drug related problem
  Interventions: Other: Detection of drug related problem in inpatient

INTERVENTIONS:
Other: Detection of drug related problem in inpatient — Detection of drug related problem in inpatient

SUMMARY:
Drug Related Problem (DRP) is defined as an event that may potentially affect the health outcomes in the patients. DRPs can occur at all stages of the medication usage process starting from prescribing to dispensing stage. Lack of follow-ups and reassessment of therapeutic outcomes may also contribute to DRPs. Pharmaceutical care is a co-operative activity in concert with other health care professionals and offered directly to the patient for improved quality use of medicines and achieving achieve the desired therapeutic outcomes. Pharmaceutical care identifies and resolves actual or potential DRPs.

DRPs pose a challenge to the clinician, and that may affect patient's clinical outcomes and may result in morbidity or mortality and increased health care costs. Health care costs may become a burden to the patient or may be to the government or to the third parties. Clinical Pharmacy is a discipline that promotes the quality use of medicines through evidence-based medicine and helps in identification and resolving DRPs. A clinical pharmacist through his/her clinical accuracy checking may identify DRPs and come out with suitable solutions to resolve the same.

Consequently, the aims of our study were to assess prevalence and characteristics of DRPs identified in inpatient and to identify factors associated with DRPs.

DETAILED DESCRIPTION:
At admission, pharmaceutics' team (senior pharmacist, one resident and two pharmacy students), conducted medication reconciliation process within 24 hours of admission or on the first working day following admission for admissions during week-ends. A medication reconciliation process was conducted according to a validated protocol. The first step consists of getting the Best Possible Medication History (BPMH), defined as the most comprehensive list of all medications taken by the patient. The second step consists of comparing the BPMH with admission prescription made by the physician in charge.

During pharmacist interview, pharmacist discussed about medication adherence and knowledge.

The third step consists of characterizing, solving and documenting DRPs. Each DRP highlighted by pharmaceutical team were collected and were classified regarding drug class and problem' types. For each patient with an identified DRP, the potential clinical impact was determined through a consensus of an expert panel: 2 pharmacists (1 hospital senior pharmacist and the resident) and 2 senior clinicians from the clinical department. The index used to rate the significance of the errors was based on the National Coordinating Council for Medication Error Reporting and Prevention (NCC MERP) Index for categorizing medication errors and adapted to get 4 severity categories with the type of error that leads to this severity: very serious, serious, moderate and minor.

For each medication, we collected its name, dosage, dosage forms and frequency of administration. For each DRP, we collected the type of DRP, the drug classes (according to anatomical therapeutic chemical classification system) and the potential clinical impact for the patient.

ELIGIBILITY:
Inclusion criteria:

- Patients aged above 18 years old, admitted to the department during the study period and hospitalized for at least 24 hours

Exclusion criteria:

- NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population was composed of patient hospitalized in Montpellier University hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2035-11-01 (Estimated); Study Completion 2036-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of drug related problems | 1 day
  Number of drug related problems identified in inpatient

SECONDARY OUTCOMES:
number of variable associated with drug related problems | 1 day
  number of variable associated with drug related problems

CONTACTS AND LOCATIONS:
Overall Officials: Cyril BREUKER, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC